CLINICAL TRIAL: NCT01548729
Title: Metabolic Efficiency of Combined Pancreatic Islet and Lung Transplant for the Treatment of End-Stage Cystic Fibrosis : a Pilot Study
Brief Title: Metabolic Efficiency of Combined Pancreatic Islet and Lung Transplant for the Treatment of End-Stage Cystic Fibrosis
Acronym: PIM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4790
Record Dates: First submitted 2012-02-10; First posted 2012-03-08 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis; Diabetes Related Cystic Fibrosis; Insulin-dependent Diabetes
Keywords: Cystic Fibrosis; Diabetes Related Cystic Fibrosis; Lung transplantation; Pancreatic islets; Insulin-dependent diabetes
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus, Type 1 | interventions — Lung Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient with cystic fibrosis (Experimental): Patients with end-stage cystic fibrosis
  Interventions: Procedure: Combined pancreatic islet and lung transplantation

INTERVENTIONS:
Procedure: Combined pancreatic islet and lung transplantation — Combined pancreatic islet and lung transplant from the same donor for the treatment of patients with end-stage cystic fibrosis

SUMMARY:
Patients with end-stage cystic fibrosis (CF) and severe CF-related diabetes (CFRD) may benefit from combined lung-pancreatic islet transplantation. A recent case series showed that combined bilateral lung and pancreatic islet transplantation is a viable therapeutic option for patients with end-stage CF and CFRD. The use of different organs from a single donor may lead to reduced immunogenicity. As the prevalence of CFRD has increased dramatically with the improved life expectancy of patients with CF, islet transplantation should be considered at the end-stage CF. By restoring metabolic control, the investigators hypothesize that islet transplantation may improve the management of CF patients undergoing lung transplant and decrease the complication rate in the early postoperative period.

ELIGIBILITY:
Inclusion criteria:

* Patient with cystic fibrosis
* Patient able to respect the protocol procedures
* Patient with end-stage respiratory insufficiency indicating a lung transplant
* Clinical history of cystic fibrosis related diabetes and/or insulin-dependent diabetes, with no residual insulin secretion (C-peptide < 0,5 ng/mL) and/or no response to IV glucagon stimulation: [peak stimulated C-peptide (T6min)/basal plasma C-peptide(T0)] < 2. The absence of insulin secretion will be verified 2 times before inclusion
* Evolution of diabetes for over 3 years
* Patient whose glycaemic control obtained with insulin therapy is not satisfactory and could significantly alter quality of life (HbA1c > 7% and/or MAGE index > 1,25). This situation is assessed by a diabetologist.
* Social Security membership or benefit from Social Welfare
* Patient who received the results of the medical evaluation required

Non-inclusion criteria:

* Patient with contra-indication for undergo a lung transplant
* Patient with an indication of heart, liver or kidney transplantation
* Patient for which poor therapeutic compliance is expected
* Patient under oral antidiabetic drug
* In women of childbearing potential: pregnancy test (urine and / or blood) positive, lactation, or unwilling to use effective contraception for the duration of the study until 3 months after the end . Men: procreation project during the study period up to 3 months after its end, or unwilling to use effective contraception patient.
* Active infection, including hepatitis B, hepatitis C, HIV
* Any history of malignancy within the past 5 years, with the exception of cutaneous basal cell carcinomas completely resected. The history of breast or melanoma cancers are an absolute contraindication
* Alcoholic intoxication or drug addiction
* Anemia (hemoglobin Hb <10g / dL in women and Hb <11 g / dL in men), lymphopenia (<1000 / uL), neutropenia (<1500 / uL) or thrombocytopenia (<100,000 / uL).
* Persistent elevated liver enzymes at baseline
* Portal hypertension identified by oesophageal varice and/or hypersplenism (platelets < 120 000 /mm3) or Child-Pugh score > 6.
* Use of a medical treatment under investigation within 4 weeks before inclusion
* All medical situation assessed by an investigator which could interfere with the good management of the project
* Patient restricted of freedom or unable to give his consent
* Patient has been included in another study that could interfere with the results of the study
* Contraindications to the use of experimental drugs (Cellcept®, prednisone, Prograf, prednisolone, methylprednisolone, and pancreatic islets)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-02-25 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Metabolic efficiency at 1 year | 1 year
  Combined criteria based on the 4 following criteria: weight increase > 5% compared to inclusion, fasting blood glucose < 1.1 g/l at 12 months post-transplant (beta score criterion), Reducing insulin requirements (expressed in UI/day) compared to inclusion & decreased in HbA1c >= 0.5% (in absolute value) compared to inclusion Success is defined by achieving at least three of these criteria

SECONDARY OUTCOMES:
Ratio [C-peptide stimulated T6min/ C-peptide basal T0] | 1 year after transplant
  Δ C peptide = [ C-peptide stimulated T6min/ C-peptide basal T0] Success if Δ C peptide > 2
Ratio [C-peptide/Glucose-Creatinine] & ratio [C-peptide/Glucose] | Every week during the first month, and every month during 1 year
HbA1c | Every 3 months during 1 year after transplant
C-peptide stimulated by glucagon | Every 3 months during 1 year after transplant
Ratio [C-peptide stimulated T6min/ C-peptide basal T0] | Every 3 months during 1 year after transplant
Microalbuminuria & proteinuria | Every 3 months during 1 year after transplant
Insulin requirements | Every month during 1 year after transplant
  Unit/day
Number of minor hypoglycemia | Every month during 1 year after transplant
  defined by a blood glucose level < 0.6g/L at which the patient is capable of self-sugaring
Number of major hypoglycemia | Every month during 1 year after transplant
Glycemic variability (MAGE) | Every 6 months during 1 year after transplant
  by continuous glycemic measurement Holter (CGMS) & glycemic reader memory analysis
duration of hypoglycemia | Every 6 months during 1 year after transplant
  by continuous glycemic measurement Holter (CGMS) & glycemic reader memory analysis
Forced Expiratory Volume (FEV1) | Every month during 1 year after transplant
Forced Vital Capacity (FVC) | Every month during 1 year after transplant
Tiffeneau-Pinelli index | Every month during 1 year after transplant
  FEV1/FVC
Nature of pulmonary infection episodes and nature of acute lung rejection if need be | Every month during 1 year after transplant
Dyspnea score according to the mMRC scale | Every month during 1 year after transplant
Oxygen saturation SaO2 room air | Every month during 1 year after transplant
Median maximum expiration flow | Every month during 1 year after transplant
Number of episodes of pulmonary rejection | Every visit during 1 year after transplant
  requiring a corticosteroid bolus
Number of days of post-transplant hospitalization and during the follow-up | Every visit during 1 year after transplant
Mortality | Every visit during 1 year after transplant
Adverse events | Every visit during 1 year after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Laurence KESSLER, MD, PhD, Principal Investigator — Hôpitaux Universitaires de Strasbourg; Pierre Yves BENHAMOU, MD, phD, Principal Investigator — University Hospital, Grenoble; Dominique Grenet, MD, Principal Investigator — HOPITAL FOCH DE SURESNES; Charles THIVOLET, MD, Principal Investigator — Hospices Civils de Lyon; Thierry BERNEY, MD PhD, Principal Investigator — CENTRE ROMAND DE TRANSPLANTATION - SUISSE
Locations (28):
- France (28):
  - CRCM AdulteCHU de Grenoble, Hôpital A. Michallon, Grenoble
  - Nephrologie, CHU Grenoble, Grenoble
  - Réanimation Cardiovasculaire et Thoracique, Hôpital Michallon, Grenoble
  - Service d'Endocrinologie, CHU de Grenoble, Grenoble
  - Service de Chirurgie Cardiaque, CHU Grenoble, Grenoble
  - Service de Radiologie Interventionnelle, CHU de Grenoble, Grenoble
  - Service de Pneumologie, Hôpital A. MICHALLON , CHU de Grenoble, Grenoble
  - Service d'Urologie et chirurgie de la Transplantation, Groupement Hospitalier Edouard Herriot, Lyon
  - Service de médecine de la transplantation et immunologie clinique, Hôpital Edouard Herriot, Lyon
  - CRCM adulte, Centre Hospitalier Lyon-Sud, Lyon
  - Service d'Endocrinologie, Pavillon médical, Lyon
  - Service d'imagerie radiologique et de médecine nucléaire, Centre Hospitalier Lyon-Sud, Lyon
  - Service de Chirurgie Thoracique, HOPITAL LOUIS PRADEL, Lyon
  - Service de pneumologie, Hôpital Louis Pradel, Lyon
  - Service de la Clinique d'Endocrinologie, maladies métaboliques et Nutrition, Nantes
  - Service de Néphrologie et Immuno-transplantation, Nantes
  - Service de Pneumologie, Nantes
  - Service de Radiologie, Nantes
  - Service d'endocrinologie, diabète et maladies métaboliques, Strasbourg
  - Service d'Anesthésie-Réanimations chirurgicales, Nouvel Hôpital Civil, Strasbourg
  - Service d'Anesthésie-Réanimations Chirurgicales, Strasbourg
  - Service de chirurgie, Nouvel Hôpital Civil, Strasbourg
  - Service de pneumologie, Nouvel Hôpital Civil, Strasbourg
  - Service de Radiologie, Hôpital de Hautepierre, Strasbourg
  - Unité d'Endocrinologie, Diabétologie et Médecine Métabolique - Hôpital Foch, Suresnes
  - Service d'Imagerie - Hôpital Foch, Suresnes
  - Service de Chirurgie Thoracique et Transplantation Pulmonaire - Hôpital Foch, Suresnes
  - Service de Pneumologie - Hôpital Foch, Suresnes

REFERENCES:
- [Derived] Rakotoarisoa L, Wagner C, Munch M, Renaud Picard B, Grenet D, Olland A, Greget M, Enescu I, Bouilloud F, Bonnette P, Guth A, Bosco D, Mercier C, Rabilloud M, Berney T, Yves Benhamou P, Massard G, Camilo C, Colin C, Arnold C, Kessler R, Kessler L; GRAGIL-TREPID Group. Feasibility and efficacy of combined pancreatic islet-lung transplantation in cystic fibrosis-related diabetes-PIM study: A multicenter phase 1-2 trial. Am J Transplant. 2022 Jul;22(7):1861-1872. doi: 10.1111/ajt.17058. Epub 2022 Apr 26. PMID 35403818